CLINICAL TRIAL: NCT05507944
Title: Fraction of Exhaled Nitric Oxide (FeNO) in an Occupational Cohort of Hairdressers
Brief Title: FeNO Hairdressers Pilot
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Bato Hammarstrøm, Senior consultant, Oslo University Hospital
Other Study IDs: 22/16786
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-08

CONDITIONS: Occupational Exposure; Environmental Exposure
Keywords: Airway irritants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare workers at Oslo University Hospital: Occupational control.
  Environmental exposure during commuting.
  Interventions: Diagnostic Test: FeNO measurement
- Hairdressers: Occupational exposure for airway irritants during hairdressing.
  Environmental exposure during commuting.
  Interventions: Diagnostic Test: FeNO measurement

INTERVENTIONS:
Diagnostic Test: FeNO measurement — Diurnal measurements before work and at 3 hours after work start.

SUMMARY:
A 5-day cohort diurnal FeNO study of exposed and unexposed to airway irritants during hair treatments and commuting.

DETAILED DESCRIPTION:
The project aims to increase the knowledge of daily variations in FeNO with emphasis on exposure of airway irritants during hairdressing treatments in an occupational setting and commuting. Daily measurements of FeNO before and after workplace exposure in an exposed and an unexposed cohort during a workweek (Monday to Saturday) will indicate patterns of proinflammatory responses in a dose-dependent manner. These may or may not be indicative of an increased risk for airway related disease. Results may be used for further studies of occupational hygiene, airway related disease and identification of endogenous volatile organic compounds during proinflammatory responses.

ELIGIBILITY:
Inclusion Criteria:

* have given informed consent.
* employed as hairdressers or at Oslo University Hospital as healthcare workers.
* scheduled work for at least 3 hours daily for 5 days in the study week.

Exclusion Criteria:

* lung disease.
* active smoker.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Employed as hairdressers or at Oslo University Hospital as healthcare workers.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Daily FeNO (ppb measured by Niox Vero) increase after occupational exposure. | 1 day.
  At start of work and after 3 hours. Hardressers vs. Health care workers.
Daily FeNO (ppb measured by Niox Vero) increase after enviromental exposure during commuting. | 1 day.
  At start of work and after 3 hours. Subgrouped after way of commuting.
Diurnal FeNO (ppb measured by Niox Vero) variations during a work week after occupational exposure. | 6 days
  At start of work and after 3 hours. Hardressers vs. Health care workers.
Diurnal FeNO (ppb measured by Niox Vero) variations during a work week after environmental exposure during commuting. | 6 days
  At start of work and after 3 hours. Subgrouped after way of commuting.

CONTACTS AND LOCATIONS:
Overall Officials: Bato Hammarstrøm, MD/PhD, Principal Investigator — Oslo University Hospital; Hilde Heiro, MD, Study Chair — Oslo University Hospital; Tonje Trulssen Hildre, MSc., Study Chair — Oslo University Hospital; Ingill Sandven, MD, Study Chair — Oslo University Hospital; Britt G Randem, MD/PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No